CLINICAL TRIAL: NCT01608139
Title: Pilot Study of Curcumin, Vorinostat, and Sorafenib in Patients With Advanced Solid Tumors
Brief Title: Study of Curcumin, Vorinostat, and Sorafenib
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sabinsa Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0574
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Advanced Solid Tumors; Curcumin; Sorafenib; Nexavar; Bay 43-9006; Vorinostat; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
MeSH Terms: interventions — Curcumin; Sorafenib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Curcumin + Sorafenib + Vorinostat (Experimental): Participant assigned to a dose level of the study drug combination based on when joined this study. Up to 9 dose levels of the study drug combination will be tested. Three (3) to 6 participants will be enrolled at each dose level of the study drug combination. During first cycle only, Curcumin initiated on Day 1, Vorinostat on Day 3 and Sorafenib on Day 5. Beginning with Cycle 1 Day 5, all agents administered continuously. Cycle of therapy is 28 days.
  Starting dose of Curcumin: 4 grams by mouth per day on Day 1. Starting dose of Sorafenib: 200 mg by mouth daily beginning on Day 5. Starting dose of Vorinostat: 100 mg by mouth daily beginning on Day 3.
  Interventions: Drug: Curcumin; Drug: Sorafenib; Drug: Vorinostat

INTERVENTIONS:
Drug: Curcumin — Starting dose: 4 grams by mouth per day. During the first cycle only, Curcumin given on Day 1. Beginning with Cycle 1 Day 5, all agents will be administered continuously.
Drug: Sorafenib — Starting dose: 200 mg by mouth daily. During the first cycle only, Sorafenib given on Day 5. Beginning with Cycle 1 Day 5, all agents will be administered continuously.
  Other Names: Nexavar; Bay 43-9006
Drug: Vorinostat — Starting dose: 100 mg by mouth daily. During the first cycle only, Vorinostat given on Day 3. Beginning with Cycle 1 Day 5, all agents will be administered continuously.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza

SUMMARY:
The goal of this clinical research study is to learn the highest tolerable dose of the combination of curcumin, vorinostat, and sorafenib that can be given to patients with advanced solid cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Curcumin is the active ingredient in the spice, turmeric. It is a natural anti-inflammatory compound and has shown anti-tumor activity in the laboratory and in clinical trials.

Vorinostat is designed to cause chemical changes in different kinds of proteins that are attached to DNA (the genetic material of cells), which may slow the growth of cancer cells or cause the cancer cells to die.

Sorafenib is designed to block the ability of important proteins to activate in cancer cells. These proteins, when active, are in part responsible for the abnormal growth and behavior of cancer cells. Blocking their activity may slow the growth of the cancer cells or cause the cancer cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of the study drug combination (curcumin, vorinostat, and sorafenib) based on when you joined this study. Up to 9 dose levels of the study drug combination will be tested.

Three (3) to 6 participants will be enrolled at each dose level of the study drug combination. The first group of participants will receive the lowest dose level of the study drug combination. Each new group will receive a higher dose of the study drug combination than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found.

The dose of the study drug combination that you receive may be lowered if you experience any intolerable side effects. You will not receive any doses of the study drug combination higher than the dose level that you are first assigned.

Study Drug Administration:

For the purposes of this study, a study drug "cycle" is 28 days long.

Starting on Day 1 of Cycle 1, you will begin taking curcumin 1 time daily.

Starting on Day 3 of Cycle 1, you will being taking vorinostat 1 time daily.

Starting on Day 5 of Cycle 1, you will begin taking sorafenib 1-2 times daily depending on the dose level you are assigned to. From this day forward, you will continue to take the study drug combination every day of each cycle.

Curcumin is a powder that comes in a paper packet, and you will take it by mouth with a full glass of water (8 oz.). Vorinostat and sorafenib are capsules that you will take by mouth. Vorinostat should be taken with food. Sorafenib should be taken without food. The capsules should be swallowed whole. You should not break, chew, or open the capsules.

Baseline Tests:

The following tests and procedures will be performed within 7 days before the first dose of the study drug combination (Day 1 of Cycle 1):

* You will have a physical exam, including measurement of your height, weight, and vital signs (blood pressure, breathing rate, heart rate, and temperature).
* You will be asked how well you are able to perform the normal activities of daily living (a performance status).
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Urine will be collected for routine tests.
* You will have an echocardiogram (ECHO) to check your heart function.
* Women who are able to become pregnant must have a negative blood (about 1 teaspoon) pregnancy test. In order to continue your participation in this study, the pregnancy test must be negative.

Study Visits:

Every week while you are receiving the study drug combination, blood (about 2 teaspoons) will be drawn for routine tests.

Before you begin each cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have an ECG.
* Urine will be collected for routine tests.
* You will be asked about any side effects you may be experiencing.

At the end of every 2 cycles (Cycles 2, 4, 6, and so on):

* You will have a chest x-ray, CT, MRI, and/or PET scan to check the status of the disease. If the study doctor thinks it is more appropriate for you, additional types of scans not listed in this consent form may need to be performed. The study doctor will discuss these scans with you, and you may be asked to sign a separate consent form that will explain the details and risks of those scans.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.

Length of Study:

You may remain on study for as long as the study doctor thinks you are benefitting from the study drugs. You will be taken off study early if the disease gets worse, you experience intolerable side effects, or the study doctor thinks it is in your best interest.

End-of-Study Visit:

Within 30 days after your last dose of the study drug combination, you will come back to the hospital for an end-of-study visit and the following tests and procedures performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* Urine will be collected for routine tests.
* You will be asked about any side effects you may be experiencing.
* If the study doctor thinks it is needed, you will have a chest x-ray, CT, MRI, and/or PET scan to check the status of the disease. If the study doctor thinks it is more appropriate for you, additional types of scans not listed in this consent form may need to be performed. The study doctor will discuss these scans with you, and you may be asked to sign a separate consent form that will explain the details and risks of those scans.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.

This is an investigational study. Curcumin is a commercially available substance, which is commonly used as a food additive. Curcumin is not FDA approved for the treatment of advanced solid cancer. At this time, curcumin is only being used in research. Vorinostat is FDA approved and commercially available for the treatment of T-cell lymphoma. Sorafenib is FDA approved and commercially available for the treatment of liver and renal cancer. At this time, the combination of curcumin, vorinostat, and sorafenib is only being used in research.

Up to 96 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an advanced solid tumor that has either failed one or more prior therapies or where there is no established standard of care therapy.
2. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 2 or better (0-2).
3. Patients must have normal organ and marrow function as defined below: Absolute neutrophil count (ANC) > 1,500/uL; Platelets > 100,000/uL; Total bilirubin within normal limits (patients with Gilbert's syndrome must have total bilirubin < 3.0 mg/dL) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x the institutional upper limit of normal (ULN); Creatinine </= 1.5 x ULN; Hemoglobin >/= 9.0 gm/dL; prothrombin time (PT)/ partial thromboplastin time (PTT) within normal limits
4. Patients must be able to understand and be willing to sign an IRB-approved written informed consent document.
5. Women of child-bearing potential (women who are not postmenopausal for at least one year or are not surgically sterile) and men must agree to use adequate contraception (e.g. barrier method) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
6. Patients must be 18 years of age or older since the safety and dosages of these study drugs has not been demonstrated in the pediatric population. However, patients who are 13 years old or older and have more than 50 kg of body weight will be eligible after consultation with their pediatric attending.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association (NYHA) Class III or IV), unstable angina pectoris, symptomatic cardiac arrhythmia, active bleeding, active thrombosis, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Inadequately controlled hypertension (defined as systolic blood pressure > 140 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications), any prior history of hypertensive crisis or hypertensive encephalopathy, and history of myocardial infarction or unstable angina within 6 months prior to study enrollment.
3. History of stroke or transient ischemic attack within 6 months prior to study enrollment and significant vascular disease (e.g., aortic aneurysm, aortic dissection) and symptomatic peripheral vascular disease.
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study. Minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
5. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or GI bleeding within 6 months prior to study enrollment; or serious, non-healing wound, ulcer, or bone fracture. Patients who have had a history of acute diverticulitis, GI obstruction, abdominal carcinomatosis, or peptic ulcer disease (known risks for bowel perforation) confirmed by endoscopy within the past 6 months, will also be excluded.
6. Patients on therapeutic warfarin with history of deep vein thrombosis and/or pulmonary embolism.
7. History of allergic reactions to the study drugs or their analogs.
8. Patients that have had any treatment specific for tumor control within 3 weeks of study drug treatment or: a. within 2 weeks if cytotoxic agents were given weekly b. within 6 weeks for nitrosoureas or mitomycin C c. within 4 half-lives for targeted agents with half lives and pharmacodynamic effects lasting less than 5 days (that includes, but is not limited to, erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents) d. failed to recover from toxic effects of any therapy prior to study entry
9. Urine for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
10. Patients with insulin dependent diabetes or poorly controlled type 2 diabetes.
11. Inability to swallow oral medication.
12. Pregnant or breastfeeding women.
13. Concurrent enrollment on another research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks
  Maximum tolerated dose (MTD) defined by dose limiting toxicities (DLTs) that occur in the first cycle. Hematological DLT defined as platelets less than 25,000/uL or bleeding associated with platelets less than 50,000/uL, ANC less than 500/uL for more than 7 days, neutropenic fever, hemoglobin less than 6.5 g/dL, or more than 14 days of delay in initiation of subsequent treatment because of inadequate hematological parameters. Nonhematological toxicities graded by using NCI CTCAE v4.0 toxicity criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson website — http://www.mdanderson.org